CLINICAL TRIAL: NCT04582357
Title: Offloaded Physical Activity Program Feasibility Assessment of Patients With Diabetic Foot Wounds
Brief Title: Physical Activity Assessment of Patients With Diabetic Foot Wounds
Acronym: EFADDIAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019_67; 2020-A02274-35 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot; Physical activity; Muscular mass; Cicatrization; Offloading
MeSH Terms: conditions — Diabetic Foot; Motor Activity; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise arm (Experimental): This arm is the only arm of the study, every patient is included in this arm, the patients will follow the physical activity program
  Interventions: Behavioral: Physical activity program

INTERVENTIONS:
Behavioral: Physical activity program — The physical activity program is a suite of several exercises which intend to improve muscular mass of targeted muscles.

SUMMARY:
The study evaluates the compliance of patients who suffer from a diabetic foot wound to follow a physical activity program, adapted to their medical condition.

This study will aslo evaluate the security of this program, and how it could improve or not the quality of life, the diabet's metabolical balance, and the wounds's cicatrization speed.

DETAILED DESCRIPTION:
The study is a prospective monocentric study, leaded in the Lille CHRU. this study is a physical activity program feasibility assessment for patients with diabetic foot wounds. The muscular mass stabilization and the physical activity is almost never used to heal diabetic feet wounds. With this study, we evaluate the compliance of patients to follow a physical activity program, which could lead to a further study, with more patients and multicentric, and it could measure the impact of this program on metabolical balance, wound size and quality of life.

The study will last 6 months, the inclusion will last 3 months, and each patient will have a 3 months follow-up time. The patient have several medical appointments in the diabetic foot unit, where the compliance will be evaluated, wound size and security will also be evaluated.

The activity program is a suite of exercises, 4 times in a week, it lasts 30 minutes?

The first day, follow-up book is given to the patient. During the follow-up, the patient will still have his usual medical appointments, which will occur at the 30th, 60th and 90th days.

Phone-call appointments will also be possible at the 15th and 45th days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Every patient over 18 years old
* Diabet whatever the type, with foot wound, whatever the size, or duration.

Exclusion Criteria:

* Medical condition : sub-gonal amputation, which makes physical activity impossible. Wound localization which would lead to a wound degradation, like the heel, the plantar face of toes.
* Administrative cause : impossibility to provide written informed consent, impossibility to be followed up during the needed duration, no medical insurance, rejection to sign the consent paper.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity program attendance | 3 months
  This outcome will evaluate the rate of patients who followed the whole physical activity program, with the help of a log book, which will be given to the patient at the first appointment

SECONDARY OUTCOMES:
Glycated hemoglobin variation | 3 months
  Evaluation of the glycated hemoglobin before inclusion and at the end of the study, to evaluate the diabet's metabolical balance
Wound size variation | 3 months
  The wound is measured with a graduated scale before inclusion and at the end of the study, the main axis is used to define the size
Quality of life variation | 3 months
  The quality of life will be measured with a simple survey before inclusion and at the end of the study, the survey is the DFS scale. the DFS evaluates the quality of life with questions like emotional impact, pain, personal satisfaction
Security | 3 months
  Patients will report any unexpected event or any injury in the log book, like hypoglycaemia or pain

CONTACTS AND LOCATIONS:
Overall Officials: Florence Baudoux, MD, Principal Investigator — University Hospital, Lille